CLINICAL TRIAL: NCT06791655
Title: Customized CAD/CAM Titanium-Milled Abutments Vs. Custom Abutments Over Immediate Implants in Class II Extraction Sockets in the Esthetic Zone: a Randomized Controlled Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMPDR042113
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Implant Therapy; Class II Extraction Sockets
Keywords: Stock abutments; Customized abutments; CAD/CAM technology; Class II extraction sockets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stock Abutment Group (Active Comparator): This group consists of 24 participants who will receive two-piece dental implants with stock abutments. This arm serves as a control group to assess the standard outcomes associated with conventional abutments used in immediate implant scenarios in the esthetic zone.
  Interventions: Device: Stock Abutment Implant
- Customized Titanium Milled Abutment Group (Experimental): This group also includes 24 participants and is considered the experimental group. These participants will receive two-piece dental implants equipped with customized cad cam titanium milled abutments. This arm is designed to evaluate the benefits of using customized abutments in terms of better soft and hard tissue integration and aesthetic outcomes compared to the standard stock abutment.
  Interventions: Device: Customized CAD CAM Titanium Milled Abutment Implant

INTERVENTIONS:
Device: Stock Abutment Implant — Participants in this intervention group receive a two-piece dental implant that utilizes a stock abutment. The stock abutment is a prefabricated component that connects the implant to the prosthetic suprastructure. This intervention aims to evaluate the standard outcomes of using stock abutments in the restoration of teeth in esthetic zones after immediate implant placement.
  Arms: Stock Abutment Group
Device: Customized CAD CAM Titanium Milled Abutment Implant — Participants in this intervention group are treated with a two-piece dental implant that includes a customized CAD CAM titanium milled abutment. These abutments are tailor-made using computer-aided design and manufacturing to fit the specific contours and needs of the patient's dental structure. This customized approach is hypothesized to offer superior integration with the soft and hard tissues, leading to better aesthetic outcomes and tissue health around the implant area.
  Arms: Customized Titanium Milled Abutment Group

SUMMARY:
Background: Immediate implant placement in esthetic zones, particularly Class II and III extraction sockets, presents challenges related to soft and hard tissue changes post-extraction. Customized abutments may offer advantages over stock abutments in managing these changes and improving clinical outcomes.

Objective: This study aims to evaluate the comparative effectiveness of customized cad cam titanium milled abutments versus stock abutments on dental implants in Class II extraction sockets in terms of soft and hard tissue integration and aesthetic outcomes.

Methods: A randomized controlled clinical and radiographic trial will be conducted at the Oral Medicine, Periodontology, Oral Diagnosis, and Radiology Department of Tanta University. Forty-eight patients requiring immediate implants in the maxillary anterior region will be randomly assigned to receive either a stock abutment or a customized titanium milled abutment. All implants will be placed using a computer-assisted surgical guide and treated with a collagen plug. Clinical and radiographic evaluations will be performed at baseline, 6 months, and 12 months, utilizing intraoral scanning and cone beam computed tomography (CBCT) to assess peri-implant mucosal levels and crestal bone thickness.

DETAILED DESCRIPTION:
Teeth loss is the worst scenario for patients as it is associated with functional, cosmetic and psychological morbidity. The most common cause of tooth loss is Periodontitis but it can also occur due to many causes as dental trauma, dental caries, developmental defects and genetic disorders.

Teeth loss not only impairs quality of life but also indirectly affects the wellbeing of the individual. The missing teeth affects the day-to-day activities of individuals like chewing, speech which results in low self-esteem, loss of confidence, less social interactions and thus hampers the work and daily activities. It may be classified as a handicapping situation Restoring missed or unrestorable teeth using dental implants in esthetic zone is a very challenging aspect of dentistry especially when aiming to restore missed teeth in esthetic zone with immediate implant as it requires a great deal of attention to place the implant finally inn a prosthetic driven position (esthetic zone is defined as the area that appears upon smiling including lip, gingiva and teeth).

While using Immediate implants in esthetic zone specially in compromised extraction sockets as classII or classIII sockets the clinicians are faced with both soft and hard tissue changes after teeth extraction , crestal and facial bone loss followed by soft tissue recession or collapse.

Peri-implant tissue health can be manifested in many items as bleeding on probing(BOP), and probing depth(PD) . In contrast to natural teeth with known reported average PD, the PD of osseointegrated successful implants are a matter of debate. Increased PD may be a sign of inflammation of peri-implant tissues. The extent to which probe penetrates is influenced by many factors such as probing force , probe diameter, roughness of the implant, inflammatory state of the periodontium, and firmness tissues around the dental implants. studies reported that successful implants allows probe penetration to approximately 3-4mm.

Many studies reported crestal bone loss after immediate implant placement as in Markus Huzeler et al who studied peri implant bone level around implants with platform switch abutments, results said that the mean values of crestal bone height at baseline were -0.09 mm +/- 0.65 mm for the platform-switched implants and -1.73 mm +/- 0.46 mm for the non -platform-switched implants.

Also in a study may by U-Covani et al that studied crestal bone changes Around implants placed into fresh extracted sockets showed that The total mean distance from implant shoulder to bone crest at 6 moths was -1.6 ± 0.32 mm.

Soft tissue changes, which are the headache after immediate implants, most of studies reported soft tissue changes after implantation in the term of mid facial gingival height and/or distal and mesial papilla. Many clinical studies revealed that approximately 20% of immediate implants suffered from mucosal recession of at least 1 mm.

In the other hand some studies reported that the type , design and shape of the abutment play an important role in both soft tissue and bone contouring .so in this study we are going to compare the use of stock abutment versus customized cad cam titanium milled abutment over dental implant to monitor the changes in both sof and hard tissue changes.

ELIGIBILITY:
Inclusion criteria:

1. Adults (20 -50)
2. Patients will be included if they have one or more of hopeless teeth without signs of acute infection in the maxillary anterior region.
3. Remaining roots or non-restorable teeth with sufficient bone apically and palatably to allow proper implant positioning with sufficient primary stability.
4. Optimal compliance as evidenced by no missed treatment appointments and a positive attitude towards oral hygiene.
5. Medically-free

Exclusion criteria:

1. Medically compromised patients and systemic conditions precluding implant and periodontal surgery.
2. Smokers, diabetics, pregnant or lactating women.

4. History of chemotherapy, radiotherapy in head and/or neck region. 5. Bisphosphonate therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Crestal Bone Thickness | Assessments were made at three points, baseline, after six months and twelve months post-implantation.
  This outcome assesses the thickness of the crestal bone around the implant. It is critical for maintaining implant stability and aesthetics, with changes potentially indicating either success in osseointegration or issues such as bone resorption.
Peri-implant Mucosal Level Changes | Assessments were made at three points, baseline, after six months and twelve months post-implantation.
  This outcome measures the changes in the peri-implant mucosal levels around the implant site, particularly looking for recession or improvement in the gum tissue adjacent to the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University., Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Robaian A, Hamed MM, Ahmed Y, Hassanein FEA. Comparative Evaluation of Customized CAD/CAM vs. Stock Titanium Abutments for Immediate Implant Placement in Class II Extraction Sockets: A Randomized Controlled Trial. Dent J (Basel). 2025 Aug 15;13(8):371. doi: 10.3390/dj13080371. PMID 40863074